CLINICAL TRIAL: NCT03578913
Title: Assessment of Peri-Implant Tissues Surrounding PEEK and Porcelain Fused to Metal Superstructures in Posterior Region (Randomized Controlled Clinical Trial)
Brief Title: PEEK Versus PFM Implant Supported Superstructure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reem Mohamed Ali Gabr, doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-06-32
Record Dates: First submitted 2018-06-24; First posted 2018-07-06 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: PEEK Implant Supported Restoration
Keywords: PFM implant supported restoration; Clinical assessment; radiographic assessment

STUDY DESIGN:
Intervention Model Description: Patient will receive a restoration with superior function, ethetic, and excellent clinical performance.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind (Patients and outcome assessors) both patient and assessor will be blinded to the assigned material. However the operator can't be blinded due to the difference in preparation and shade of the ceramic materials. Reem Gabr will be responsible for the try-in and final delivery of the crowns.
  -The assessor will assess all outcomes blinded to the material assigned for each patient.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- porcelain fused to metal crown (Active Comparator): Although metal free restorations are gained popularity recently, PFM restorations, whether they are tooth-supported or implant-supported are still considered as the gold standard due to their excellent biocompatibility, consistent esthetics, superior strength, and marginal adaptation.2 PFM restorations are also considered durable and long-lasting
  Interventions: Other: PEEK crown; Other: PFM Crown
- PEEK crown (Experimental): The main concern of dental implants is their lack of elasticity, therefore with the use of PFM, all ceramic or zirconia crowns; the load is directly transferred to bone. That is why up till now researchers are in quest of different materials to enhance soft and hard tissue reaction around implant supported restorations. Recently the use of PEEK as a final restoration on dental implants has wide acceptance, due to its excellent biocompatibility and exceptional physical and chemical properties regarding toughness, hardness and elasticity. In term of load cushioning capacity of the prosthetic elements, PEEK has a comparable modulus of elasticity (4GPa) to that of bone (4.2GPa). Thus, the bone could allow bone stimulation favoring its remodeling without overloading
  Interventions: Other: PEEK crown; Other: PFM Crown

INTERVENTIONS:
Other: PEEK crown — The main concern of dental implants is their lack of elasticity, therefore with the use of PFM, all ceramic or zirconia crowns; the load is directly transferred to bone. That is why up till now researchers are in quest of different materials to enhance soft and hard tissue reaction around implant supported restorations. Recently the use of PEEK as a final restoration on dental implants has wide acceptance, due to its excellent biocompatibility and exceptional physical and chemical properties regarding toughness, hardness and elasticity. In term of load cushioning capacity of the prosthetic elements, PEEK has a comparable modulus of elasticity (4GPa) to that of bone (4.2GPa). Thus, the bone could allow bone stimulation favoring its remodeling without overloading.
  Other Names: polyetherether ketone
Other: PFM Crown — Although metal free restorations are gained popularity recently, PFM restorations, whether they are tooth-supported or implant-supported are still considered as the gold standard due to their excellent biocompatibility, consistent esthetics, superior strength, and marginal adaptation.2 PFM restorations are also considered durable and long-lasting
  Other Names: metal ceramic restoration

SUMMARY:
The purpose of this study is to evaluate the influence of two superstructure materials Porcelain Fused to Metal (PFM) and PEEK on peri- implant soft and hard tissue reaction clinically.

DETAILED DESCRIPTION:
Nowadays the use of dental implants for restoring missing teeth has gained a wide acceptance, due to its high success rate.

Dental implants differ from natural teeth in transmission of functional loads to the bone, where natural teeth and their periodontal ligaments provide proprioception, early detection of occlusal loads and have a shock-absorbing function. Sensitivity and mobility of natural teeth cannot be duplicated in osseointegrated implants,1 therefore most of the forces are concentrated at the crest of the ridge leading to different living reaction including bone resorption and subsequent implant loss.

Minimizing the occlusal loads on osseointegrated implants through selection of a new superstructure material that can absorb part of this excessive force could be believed to be a determining factor in the long-term success of an implant treatment program.

Many restorative materials are used nowadays for construction of final restoration of implant supported superstructures including porcelain fused to metal (PFM), all ceramic, zirconia, hybrid ceramics, and polyetheretherketone (PEEK). PFM restorations are still considered as the gold standard because of their excellent biocompatibility, consistent esthetics, superior strength, and marginal adaptation. Recently, the use of new resilient superstructure material like PEEK-based restoration on implant prosthetics could modify the occlusal forces with subsequent cushioning during function.

ELIGIBILITY:
Inclusion criteria:

* Patients above 18 years old.
* Patients able to read and sign the informed consent document.
* Medically free patients or with controlled systemic disease.
* Patients with good bone quality and quantity.
* Patients willing to return for follow-up examinations and evaluation.
* Patients having single successfully osseointegrated implant in posterior region.

Exclusion criteria

* Young patients in growth stage.
* Patients with unsuitable implantation sites (patients with major boney defects or sever bone resorption)
* Pregnant women to avoid any complication that may occur in dental office.
* Patients with uncontrolled systemic disease (hypertensive patient or uncontrolled diabetic patient)
* Psychiatric problems or unrealistic expectations.
* Multiple adjacent missing teeth.
* Patients with bad oral hygiene.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scales (VAS) for measuring the patient satisfaction | 12 months
  Visual analogue scales will be used before the treatment and at the follow-ups to record and evaluate subjective patient's perceptions including the appraisal of function eating, esthetics, sense, speech, and self-esteem. The patients were asked to mark their subjective perception in each category on a horizontal line (100 mm in length), 1 mm (the minimum score) corresponded to 1% of satisfaction and 100 mm (the maximum score) corresponded to 100% of satisfaction.

SECONDARY OUTCOMES:
Crestal bone loss | 12 months
  Intraoral X-rays will be made using the long-cone parallel technique for the two groups. All radiographs were digitized for evaluation of the bone levels (BL) at different time points. The marginal BL was determined by measuring the distance between the implant shoulder (reference) and the most coronal bone-to implant contact. These measurements were made by two independent examiners mesially and distally of the implants and in 0.1-mm increments
Gingival index | 12 months
  Gingival index of the two groups will be assessed by the Loe & Silness gingival index as follow:
  * Grade 0: (Normal gingival) Natural coral pink gingival.
  * Grade 1: (Mild inflammation) Slight change in color, slight edema. No bleeding on probing.
  * Grade 2: (Moderate inflammation) Redness, edema and glazing. Bleeding on probing.
  * Grade 3: (Severe inflammation) Marked redness and edema. Tendency to spontaneous bleeding. Ulceration.
bleeding index | 12 months
  Bleeding index of the two groups will be assessed by Modified sulcus bleeding index11 With a periodontal probe (PCB 12; Hu-Friedy, Leimen, Germany) inserted about 1mm into the peri-implant epithelium, the sulcus was scratched over its facial and oral surface as follow:
  * Grade 0: No bleeding.
  * Grade 1: Isolated points of bleeding.
  * Grade 2: The blood forms a confluence line at the epithelium.
  * Grade 3: Massive bleeding/spontaneous bleeding.
Probing depth | 12 months
  Probing pocket depth (PPD) for the two groups will be measured from the mucosal margin to the bottom of the probeable pocket in millimeters with a periodontal probe (PCB 12; Hu-Friedy, Leimen, Germany) at four aspects per implant
  * mesial
  * distal
  * buccal
  * lingual The subscales will be summed and an average will be taken.

REFERENCES:
- [Background] Weinberg LA. The biomechanics of force distribution in implant-supported prostheses. Int J Oral Maxillofac Implants. 1993;8(1):19-31. PMID 8468083
- [Background] Walton TR. An up to 15-year longitudinal study of 515 metal-ceramic FPDs: Part 1. Outcome. Int J Prosthodont. 2002 Sep-Oct;15(5):439-45. PMID 12375457
- [Background] Ponnappan RK, Serhan H, Zarda B, Patel R, Albert T, Vaccaro AR. Biomechanical evaluation and comparison of polyetheretherketone rod system to traditional titanium rod fixation. Spine J. 2009 Mar;9(3):263-7. doi: 10.1016/j.spinee.2008.08.002. Epub 2008 Oct 1. PMID 18838341
- [Background] Han KH, Lee JY, Shin SW. Implant- and Tooth-Supported Fixed Prostheses Using a High-Performance Polymer (Pekkton) Framework. Int J Prosthodont. 2016 Sep-Oct;29(5):451-4. doi: 10.11607/ijp.4688. PMID 27611747
- [Background] Parmigiani-Izquierdo JM, Cabana-Munoz ME, Merino JJ, Sanchez-Perez A. Zirconia implants and peek restorations for the replacement of upper molars. Int J Implant Dent. 2017 Dec;3(1):5. doi: 10.1186/s40729-016-0062-2. Epub 2017 Feb 20. PMID 28220366
- [Background] Mombelli A, Marxer M, Gaberthuel T, Grunder U, Lang NP. The microbiota of osseointegrated implants in patients with a history of periodontal disease. J Clin Periodontol. 1995 Feb;22(2):124-30. doi: 10.1111/j.1600-051x.1995.tb00123.x. PMID 7775668
- [Background] Landry RG, Jean M. Periodontal Screening and Recording (PSR) Index: precursors, utility and limitations in a clinical setting. Int Dent J. 2002 Feb;52(1):35-40. doi: 10.1111/j.1875-595x.2002.tb00595.x. PMID 11931220
- [Background] UPDEGRAVE WJ. The paralleling extension-cone technique in intraoral dental radiography. Oral Surg Oral Med Oral Pathol. 1951 Oct;4(10):1250-61. doi: 10.1016/0030-4220(51)90084-9. No abstract available. PMID 14882798